CLINICAL TRIAL: NCT01648686
Title: Bone Healing After Dental Extraction in Postmenopausal Osteoporotic Women Treated With Alendronate Per os (70 mg Weekly)
Brief Title: Bone Healing After Dental Extraction in Postmenopausal Osteoporotic Women Treated With Alendronate Per os Weekly
Acronym: BOCOMEDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P110126
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Alveolar Bone Healing After Dental Extraction
Keywords: Alendronate; Dental extraction; Bone healing; postmenopausal women; dental radiography
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women treated by bisphosphonate (Active Comparator): Postmenopausal osteoporotic women treated by alendronate 70 mg weekly per os
  Interventions: Procedure: Dental extraction
- Women didn't treat by bisphosphonate (Sham Comparator): Postmenopausal osteoporotic women untreated by bisphosphonates
  Interventions: Procedure: Dental extraction

INTERVENTIONS:
Procedure: Dental extraction — 3 dental radiographies realised immediately, then 30 days, then 90 days after dental extraction

SUMMARY:
The purpose of this study is to determine whether the oral alendronate treatment of post-menopausal osteoporosis could be a risk factor for jaw bone healing after dental extraction.

DETAILED DESCRIPTION:
Alendronate is the main oral bisphosphonate used in the treatment and the prevention of the postmenopausal osteoporosis because of its high antiresorbant ability for bone tissue. Alendronate delayed bone healing after dental extraction on animals models, murine as canine. Anti-angiogenic and anti-osteoclastic characteristics are suggested to explain this phenomenon. There is no available data in human and it is now well known that bisphosphonates are involved in the occurrence of osteonecrosis of the jaws even if this major adverse effect seems to be very seldom with oral alendronate. Moreover, bisphosphonate showed toxicity for oral mucosal cells. The main aim of this study is to quantify the impact of oral alendronate weekly treatment on bone and mucosa healing after dental extraction in postmenopausal osteoporotic women. A secondary aim is to investigate a panel of 50 peptids potentially involved in bone and mucosal healing and to detect changes in their rates by salivary proteomic approach. The investigators hope so identify salivary biomarkers of bone and/or mucosa healing in these women.

Our hypothesis is that after dental extraction, bone healing could be delayed in postmenopausal osteoporotic women treated with oral weekly alendronate (BP+ group) versus matched osteoporotic women untreated with bisphosphonates (BP- group).

This is a prospective and multicentric (17 investigation centers dispatched in France) study including 140 osteoporotic postmenopausal women treated weekly with oral bisphosphonates (BP+ group) and 140 osteoporotic postmenopausal women untreated with bisphosphonates (BP- group). This is a clinical follow-up study (T0, T0 + 7, T0 + 30, T0 + 90 days), a radiological study (T0, T0 + 30, T0 + 90 days), and a salivary proteomic study (T0, T0 + 30, T0 + 90 days). This is a 4 years study starting in april 2012 (anticipated date).

The main investigated parameters are:

* Bone healing: Bone filling rate (in %) of the post-extractional alveolar socket (BFR) at T0, T0 + 30 and T0 + 90 days by a radiographic approach.
* Mucosa healing: mucosal injury by metric approach at T0 and T0 + 30 days.
* Salivary biomarkers: Fifty peptides by proteomic approach at T0 and T0 + 30 days;

The investigators expect that this study will allow us to build a reference scale of bone and mucosa healing in osteoporotic postmenopausal women treated weekly by oral alendronate. This scale will be a helpful tool for dental physicians. The investigators hope also to identify salivary biomarkers variations to make a diagnosis and a prognosis tool of worse bone healing in these patients.

Perspectives of this study is to constitute a national network of deleterious effect on bone healing in such women patients and to up-date guidelines in this area.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporotic women
* Treated with alendronate per os (70 pg weekly) for BP+ experimental group and untreated with this therapy for the BP
* Control group
* Subjected to single root tooth extraction- 45 to 70 years of age

Exclusion Criteria:

* Maxillofacial irradiations
* Dental extraction with adjunction of material interfering with bone healing
* Severe pathologies inconsistent with this study
* Bisphosphonate treatment for BP- control group
* Women treated with denosumab (prolia®)
* Women already included to an another dental extraction

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Alveolar socket filled by new bone | 3 months after extraction
  Rate in % of the alveolar socket filled by new bone

SECONDARY OUTCOMES:
Mucosal injury | 7 days after extraction
  Direct measure of mucosal injury wtih a mini-electronic caliper

CONTACTS AND LOCATIONS:
Overall Officials: Christian ROUX, MD, PhD, Study Chair — Hôpital Cochin
Locations (1):
- Hotel-Dieu Hospital, Nantes, France

REFERENCES:
- [Background] Lesclous P, Cloitre A, Catros S, Devoize L, Louvet B, Chatel C, Foissac F, Roux C. Alendronate or Zoledronic acid do not impair wound healing after tooth extraction in postmenopausal women with osteoporosis. Bone. 2020 Aug;137:115412. doi: 10.1016/j.bone.2020.115412. Epub 2020 May 20. PMID 32404281